CLINICAL TRIAL: NCT03754413
Title: A Multicenter Randomized, Evaluator-Blinded, "No Treatment" Controlled Study to Evaluate the Effectiveness and Safety of Neuramis® Volume Lidocaine for Volume Augmentation in the Mid-Face
Brief Title: Neuramis® Volume Lidocaine for Volume Augmentation in the Mid-Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MT08-CN16MFV702
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Mid Face Volume Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational medical device (Experimental): Neuramis® Volume Lidocaine
  Interventions: Device: experimental
- Comparator device (Other): No-treatment
  Interventions: Drug: comparator

INTERVENTIONS:
Device: experimental — Neuramis® Deep Lidocaine
  Arms: Investigational medical device
Drug: comparator — No-treatment
  Arms: Comparator device

SUMMARY:
To evaluate the effectiveness and safety of Neuramis® Volume Lidocaine for volume augmentation in the mid-face.

DETAILED DESCRIPTION:
This is a multicenter, randomized, evaluator-blinded, "no-treatment" controlled study conducted in normal, healthy subjects. This study is anticipated to enroll approximately 236 male and/or female subjects between the ages of 20 to 75 years, inclusive, who desire volume augmentation to correct deficit in their mid-face volume.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 20 to 75 years of age
2. Subjects who desire volume augmentation to correct deficit in the mid-face volume that is rated as Grade 3, 4, or 5 on the Facial Volume Scale

Exclusion Criteria:

1. Subjects who have received anti coagulation, anti-platelet, or thrombolytic medications, anti-inflammatory drugs.
2. Subjects who have undergone facial plastic surgery in the face area below the level of the lower orbital rim, tissue grafting, or tissue augmentation with silicone, fat, or other permanent, or semi-permanent dermal fillers or are planning to undergo any of these procedures at any time during the clinical investigation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Total Facial Volume Scale(FVS) improvement rate at Week 24 | Week 24
  Facial Volume Scale score ranges from 0-5 with higher score indicating increasing severity of mid-face volume deficit / Proportion of subjects with Facial Volume Scale(FVS) showing ≥1-point improvement (Facial Volume Scale decrease ≥1) at Week 24 compared to Baseline

SECONDARY OUTCOMES:
6-point Facial Volume Scale(FVS) improvement rate at Weeks 4, 12, 36, and 52 | Weeks 4, 12, 36, and 52
  The proportion of subjects with 6-point Facial Volume Scale(FVS) decrease ≥1 from Baseline as assessed at Weeks 4, 12, 36, and 52.
Change in 6-point Facial Volume Scale(FVS) at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  Change in 6-point Facial Volume Scale(FVS) at Weeks 4, 12, 24, 36, and 52
Global Aesthetic Improvement Scale(GAIS) improvement rate at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  Global Aesthetic Improvement Scale(GAIS) improvement rate is defined as the proportion of subjects with GAIS score ≤3

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hopsital, Beijing, China